CLINICAL TRIAL: NCT03510741
Title: A Multicentre 12-week Randomised Double-blind Placebo Controlled Feasibility Trial of Sodium Benzoate and/or N-acetylcysteine Added to TAU in Patients With Early Schizophrenia Spectrum Disorder.
Brief Title: Sodium Benzoate and/or N-Acetylcysteine Added to TAU in Patients With Early Schizophrenia Spectrum Disorder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: PILL-Sodium Benzoate & NAC-001
Record Dates: First submitted 2018-04-04; First posted 2018-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia; Schizophreniform Disorders; Schizoaffective Disorder
Keywords: Schizophrenia; Sodium Benzoate; N-Acetylcysteine; NMDA receptor; Psychopharmacology; Anti-oxidant; Inflammation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Inflammation | interventions — Sodium Benzoate; Acetylcysteine

STUDY DESIGN:
Intervention Model Description: This will be a 2x2 factorial design trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind placebo controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sodium Benzoate (Active Comparator): Sodium Benzoate added to TAU will be administered at 1000mg daily
  Interventions: Drug: Sodium Benzoate
- N-Acetylcysteine (Active Comparator): N-Acetylcysteine added to TAU 1000 mgs twice daily dose
  Interventions: Drug: N-Acetylcysteine
- Placebo (Active Comparator): Placebo added to TAU
  Interventions: Drug: Placebo
- Sodium Benzoate Plus N-Acetylcysteine (Active Comparator): Sodium Benzoate will be administered at 1000mg daily and NAC 1000 mgs twice daily dose
  Interventions: Drug: Sodium Benzoate Plus N-Acetylcysteine

INTERVENTIONS:
Drug: Sodium Benzoate — Sodium Benzoate will be administered at 1000mg daily
  Arms: Sodium Benzoate
Drug: N-Acetylcysteine — N-Acetylcysteine 1000 mgs twice daily dose
  Arms: N-Acetylcysteine
Drug: Placebo — Placebo added to TAU
  Arms: Placebo
Drug: Sodium Benzoate Plus N-Acetylcysteine — Sodium Benzoate will be administered at 1000mg daily and NAC 1000 mgs twice daily dose
  Arms: Sodium Benzoate Plus N-Acetylcysteine

SUMMARY:
This study aims to determine if the addition of Sodium Benzoate and / or NAC to TAU will be acceptable and tolerable and result in overall improvement of symptoms, social and cognitive functioning in patients with early schizophrenia spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female patients aged between 18-35 years.
2. Diagnosis of schizophrenia confirmed by SCID interview meeting DSM-V criteria for schizophrenia, schizophreniform or schizoaffective psychosis.
3. Stable on medication for the past four weeks
4. In contact with mental health services
5. Within 5 years of diagnosis of psychotic illness
6. Able to demonstrate the capacity to provide informed consent as assessed by their own clinician
7. Able to complete the required evaluations and take oral medication.
8. Effective contraceptive precautions (either the use of barrier methods or the oral contraceptive pill) to be taken by women of child-bearing age. A negative pregnancy test will be required in order to meet inclusion criteria.

Exclusion Criteria:

1. Prior history of intolerance or serious side effects to Sodium Benzoate or N-acetylcystine.
2. Concomitant use of Ascorbic acid
3. Active substance abuse (except nicotine or caffeine) or dependence within the last three months according to DSM-V criteria.
4. Relevant CNS or other medical disorders.
5. Pregnant or breast feeding
6. Diagnosis of Moderate to Severe Learning Disability
7. Relevant current or past haematological, hepatic, renal, neurological or other medical disorder in the opinion of the principal investigator (PI) or the responsible clinician, that may interfere with the trial.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention ( including recruitment rates and drop outs) | Recruitment within 12 months of study start start date
  Feasibility estimates of delivering the intervention including recruitment rates and drop outs

SECONDARY OUTCOMES:
Overall improvement in symptoms using the Positive and Negative Syndrome Scale (PANSS) total score | change in scores from Baseline to 12 weeks
  The PANSS is measured on a 7-point scale, and is a 30-item structured clinical interview assessing symptom severity over the previous week. The PANSS scale has a maximum score of 210 and a minimum of 30. Higher scores indicate higher severity of illness.

OTHER OUTCOMES:
Improvement in positive and/or negative symptoms subscales measured using the PANSS. | change in scores from Baseline to 12 weeks
  The PANSS is measured on a 7-point scale, and is a 30-item structured clinical interview assessing symptom severity over the previous week. The PANSS scale has a maximum score of 210 and a minimum of 30. Higher scores indicate higher severity of illness.
Improvement on Clinical Global Impression (CGI) Scale and Social and Occupational Functioning Assessment (SOFA) scales. | change in scores from Baseline to 12 weeks
  Clinical Global Impression (CGI) Scale is an observer rated clinical severity measure. The minimum score is 1 and maximum 7. Higher scores indicate severity of illness. Social and Occupational Functioning Assessment (SOFA) scale is a measure of current functioning, with scores ranging from 0 to 100. Higher scores represent higher functioning
Improvement in cognitive functioning as measured using CogState Schizophrenia Battery. | change in scores from Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Imran B Chaudhry, MD, Principal Investigator — Ziauddin Hospital
Locations (5):
- Pakistan (5):
  - Balochistan Institute of Behavioral Science, Quetta, Balochistan
  - Institute of Psychiatry, Rawalpindi, Rawalpindi, Islamabad
  - Abbasi Shaheed Hsopital, Karachi, Sindh
  - Civil Hospital Karachi, Karachi, Sindh
  - Karwan e Hayat, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berk M, Copolov D, Dean O, Lu K, Jeavons S, Schapkaitz I, Anderson-Hunt M, Judd F, Katz F, Katz P, Ording-Jespersen S, Little J, Conus P, Cuenod M, Do KQ, Bush AI. N-acetyl cysteine as a glutathione precursor for schizophrenia--a double-blind, randomized, placebo-controlled trial. Biol Psychiatry. 2008 Sep 1;64(5):361-8. doi: 10.1016/j.biopsych.2008.03.004. Epub 2008 Apr 23. PMID 18436195
- [Background] Chaudhry IB, Husain N, Drake R, Dunn G, Husain MO, Kazmi A, Hamirani MM, Rahman R, Stirling J, Deakin W. Add-on clinical effects of simvastatin and ondansetron in patients with schizophrenia stabilized on antipsychotic treatment: pilot study. Ther Adv Psychopharmacol. 2014 Jun;4(3):110-6. doi: 10.1177/2045125313511487. PMID 25057343
- [Background] Farokhnia M, Azarkolah A, Adinehfar F, Khodaie-Ardakani MR, Hosseini SM, Yekehtaz H, Tabrizi M, Rezaei F, Salehi B, Sadeghi SM, Moghadam M, Gharibi F, Mirshafiee O, Akhondzadeh S. N-acetylcysteine as an adjunct to risperidone for treatment of negative symptoms in patients with chronic schizophrenia: a randomized, double-blind, placebo-controlled study. Clin Neuropharmacol. 2013 Nov-Dec;36(6):185-92. doi: 10.1097/WNF.0000000000000001. PMID 24201233
- [Background] Lane HY, Lin CH, Green MF, Hellemann G, Huang CC, Chen PW, Tun R, Chang YC, Tsai GE. Add-on treatment of benzoate for schizophrenia: a randomized, double-blind, placebo-controlled trial of D-amino acid oxidase inhibitor. JAMA Psychiatry. 2013 Dec;70(12):1267-75. doi: 10.1001/jamapsychiatry.2013.2159. PMID 24089054
- [Background] Lin CH, Lin CH, Chang YC, Huang YJ, Chen PW, Yang HT, Lane HY. Sodium Benzoate, a D-Amino Acid Oxidase Inhibitor, Added to Clozapine for the Treatment of Schizophrenia: A Randomized, Double-Blind, Placebo-Controlled Trial. Biol Psychiatry. 2018 Sep 15;84(6):422-432. doi: 10.1016/j.biopsych.2017.12.006. Epub 2017 Dec 26. PMID 29397899
- [Background] Chaudhry IB, Hallak J, Husain N, Minhas F, Stirling J, Richardson P, Dursun S, Dunn G, Deakin B. Minocycline benefits negative symptoms in early schizophrenia: a randomised double-blind placebo-controlled clinical trial in patients on standard treatment. J Psychopharmacol. 2012 Sep;26(9):1185-93. doi: 10.1177/0269881112444941. Epub 2012 Apr 23. PMID 22526685
- [Derived] Husain MO, Chaudhry IB, Khoso AB, Husain MI, Ansari MA, Mehmood N, Naqvi HA, Nizami AT, Talib U, Rajput AH, Bassett P, Foussias G, Deakin B, Husain N. Add-on Sodium Benzoate and N-Acetylcysteine in Patients With Early Schizophrenia Spectrum Disorder: A Multicenter, Double-Blind, Randomized Placebo-Controlled Feasibility Trial. Schizophr Bull Open. 2024 Feb 9;5(1):sgae004. doi: 10.1093/schizbullopen/sgae004. eCollection 2024 Jan. PMID 39144112